CLINICAL TRIAL: NCT07035431
Title: A Prospective Multicenter Trial Evaluating the Safety and Effectiveness of Endo-SPONGE for the Treatment of Anastomotic or Hartmann's Stump Leakages in the Lower Pelvic Area
Brief Title: Endo-SPONGE for Treatment of Anastomotic or Hartmann's Stump Leakages in Lower Pelvic Area
Acronym: DRAIN Lower
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7212
Record Dates: First submitted 2025-06-10; First posted 2025-06-25 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Anastomotic Leaks; Hartmanns Stump Leakage
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Endoscopic Vacuum Therapy (EVT) Device (Experimental)
  Interventions: Device: Endo-SPONGE

INTERVENTIONS:
Device: Endo-SPONGE — The intervention involves the placement of an Endo-SPONGE in the leakage cavity, and applying suction to facilitate drainage.

SUMMARY:
This study is intended to evaluate the safety and effectiveness of Sponge-based Endoscopic Vacuum Therapy (EVT) using Endo-SPONGE for the treatment of Anastomotic Leaks (AL) or Hartmann's stump leakages following colorectal surgery in a prospective multi-center study.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed grade B anastomotic leak as per the ISGRC (International Study Group of Rectal Cancer) grading system after colorectal surgery.
* Subject is eligible for endoscopic intervention.
* Subject has a transmural defect of at least 2 cm in diameter following colorectal surgery in the lower pelvic area.
* Subject has an anastomotic or Hartmann's stump leak located within an extraperitoneal cavity.
* Subject has pre-existing diverting ostomy or an ostomy created prior to the first Endo-SPONGE placement.
* Subject understands the trial requirements and is willing and able to comply with the study procedures, all protocol-required follow up evaluations and provide written informed consent to participate in the study.
* Investigator decision that EVT is the most suitable treatment of the available treatment options.

Exclusion Criteria:

* Subject is under 18 years of age.
* Potentially vulnerable subject, including, but not limited to pregnant women.
* Subject has undergone EVT or other similar interventions for the current colorectal indication.
* Subject had colorectal surgery more than 60 days prior to the planned study procedure.
* Subject has any necrotic tissue that would require endoscopic debridement prior to Endo-SPONGE placement.
* Subject has known contraindication for EVT as per the IB.
* Subject is currently enrolled in another investigational study that would directly interfere with the current study, without prior written approval from the sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events | Day 0 Study Procedure to end of study; up to 6 months
  The proportion of subjects with one or more study device or endoscopic or study procedure-related Serious Adverse Events (SAEs) occurring up to 3 months after the last study device removal.
Clinical Success | Day 0 Study Procedure to the last study device removal; up to 3 months
  The proportion of subjects that demonstrate clinical success, which is defined as closure of the anastomotic or Hartmann's stump leak, confirmed via endoscopy or contrast-enhanced computed tomography imaging within 3 months after the study procedure without the need for an additional endoscopic or surgical intervention.

SECONDARY OUTCOMES:
Technical Success | Day 0 Study Procedure to the last study device exchange; up to 3 months
  Defined as the ability to deploy the Endo-SPONGE in the intended location. This will be calculated for study procedure and every Endo-SPONGE Exchange that is attempted.
Closure Time | Day 0 Study Procedure to the last study device removal; up to 3 months
  Time to colorectal anastomotic or Hartmann's stump leak closure.
Rate of Reinterventions | From last study device removal to end of study; 3 months
  Rate of Reinterventions after closure of the anastomotic or Hartmann's stump leak.
Time to Additional Intervention | Day 0 Study Procedure to the last study device removal; up to 3 months
  Time to additional intervention, if Endo-SPONGE treatment is insufficient.
Leak Recurrence | From last study device removal to end of study; 3 months
  Leak recurrence within 3 months following completion of Endo-SPONGE therapy.
Endo-SPONGE Exchanges | Day 0 Study Procedure to last study device removal; up to 3 months
  Number of Endo-SPONGE exchanges needed to reach clinical success.
Length of Hospitalization | Day 0 Study Procedure to end of study; up to 6 months
  Length of Hospitalization.
Mortality Rate | Day 0 Study Procedure to end of study; up to 6 months
  Mortality rate through 3-month follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Pauli, MD, Principal Investigator — Penn State Health
Locations (8):
- United States (8):
  - Barnes Jewish Hospital, St Louis, Missouri
  - Mount Sinai, New York, New York
  - New York Presbyterian / Columbia University Irving Medical Center, New York, New York
  - Ohio State University Medical Center, Columbus, Ohio
  - Penn State Health, Hershey, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - University of Washington Medical Center, Seattle, Washington
  - Marshall University Medical Center, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No